CLINICAL TRIAL: NCT01460329
Title: Comparing Cardiac Output Measurements in Critically Ill Children Using Ultrasonic Cardiac Output Monitor and Transthoracic Echocardiography.
Brief Title: Comparing Cardiac Output Measurements in Critically Ill Children Using USCOM and Transthoracic ECHO
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Principal Investigator, Nina Verdino, MD, Principal Investigator, University of North Carolina, Chapel Hill
Other Study IDs: 11-1178
Record Dates: First submitted 2011-10-24; First posted 2011-10-26 (Estimated); Last update posted 2013-05-06 (Estimated); Status verified 2013-05

CONDITIONS: Critical Illness; Pediatrics
Keywords: intensive care units; pediatric; cardiac index; Doppler Ultrasonography
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- USCOM Cardiac index
  Interventions: Device: Ultrasonic Cardiac Output Monitor (USCOM).

INTERVENTIONS:
Device: Ultrasonic Cardiac Output Monitor (USCOM). — This device is FDA approved and based on the principles of ECHO using continuous-wave Doppler ultrasound to measure cardiac output.
  Other Names: USCOM

SUMMARY:
The purpose of this study is to compare the accuracy and precision of two non-invasive methods of measuring cardiac output in critically ill children (<18 yrs). The participants will include any patient admitted to Pediatric intensive care unit (PICU) requiring a trans-thoracic ECHO (TTE) as part of their treatment plan. Measurements of intermittent cardiac output will be obtained and compared on participants using standard 2-D TTE and Ultrasound Cardiac Output Monitor (USCOM).

ELIGIBILITY:
Inclusion Criteria:

* Any UNC PICU patient <18 yrs requiring a transthoracic ECHO (TTE) as standard of care.
* Gestational age >36 weeks
* Wt > 2 kg
* Written informed parental permission

Exclusion Criteria:

* Any patient with known unrepaired intracardiac shunt lesion (ASD,PDA,VSD)
* any post operative patient with delayed closure of chest
* parental refusal to participate

Ages: 1 Day to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The subjects for this study can be either male or female and not limited by race or ethnicity. They will include critically ill pediatric patients, less than 18 yrs of age, being treated in the Pediatric intensive care unit.
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2011-10; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Cardiac Index | measured at the time of study

CONTACTS AND LOCATIONS:
Overall Officials: Nina J Verdino, MD, Principal Investigator — East Carolina University; Keith C Kocis, MD, Study Chair — University of North Carolina, Chapel Hill
Locations (1):
- UNC Children's Hospital, Chapel Hill, North Carolina, United States